CLINICAL TRIAL: NCT05987332
Title: IDE196 (Darovasertib) in Combination With Crizotinib Versus Investigator's Choice of Treatment as First-line Therapy in HLA-A2 Negative Metastatic Uveal Melanoma (DAR-UM-2)
Brief Title: IDE196 (Darovasertib) in Combination With Crizotinib as First-line Therapy in Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDE196-002
Record Dates: First submitted 2023-07-12; First posted 2023-08-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Uveal Melanoma
Keywords: IDE196; Darovasertib; Protein Kinase C; Metastatic Uveal Melanoma; Melanoma; Ocular Oncology; Ophthalmology; Crizotinib; Ocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Crizotinib; pembrolizumab; Ipilimumab; Nivolumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2a Dose Optimization of IDE196 + crizotinib (Experimental): Multiple doses of IDE196 will be tested in combination with fixed dose of crizotinib to identify the optimal combination dose.
  Interventions: Drug: IDE196; Drug: Crizotinib
- Phase 2b / 3 Chosen Combination dose of IDE196 + crizotinib (Experimental): Chosen combination dose of IDE196 + crizotinib will be tested in additional participants.
  Interventions: Drug: IDE196; Drug: Crizotinib
- Phase 2a / 2b / 3 Comparator Arm (Active Comparator): Participants will receive investigator's choice of Pembrolizumab, Ipilimumab + Nivolumab, or Dacarbazine.
  Interventions: Drug: Pembrolizumab; Drug: Ipilimumab; Drug: Nivolumab; Drug: Dacarbazine

INTERVENTIONS:
Drug: IDE196 — Dosed orally, twice daily
  Other Names: Darovasertib
  Arms: Phase 2a Dose Optimization of IDE196 + crizotinib; Phase 2b / 3 Chosen Combination dose of IDE196 + crizotinib
Drug: Crizotinib — Dosed orally, twice daily
  Other Names: XALKORI
  Arms: Phase 2a Dose Optimization of IDE196 + crizotinib; Phase 2b / 3 Chosen Combination dose of IDE196 + crizotinib
Drug: Pembrolizumab — IV administration every 3 weeks
  Other Names: Keytruda
  Arms: Phase 2a / 2b / 3 Comparator Arm
Drug: Ipilimumab — IV administration every 3 weeks for 4 Cycles
  Other Names: Yervoy
  Arms: Phase 2a / 2b / 3 Comparator Arm
Drug: Nivolumab — IV administration every 3 Weeks for 4 Cycles, thereafter every 4 Weeks maintenance
  Other Names: Opdivo
  Arms: Phase 2a / 2b / 3 Comparator Arm
Drug: Dacarbazine — IV administration every 3 Weeks
  Other Names: DTIC-Dome
  Arms: Phase 2a / 2b / 3 Comparator Arm

SUMMARY:
This is a Phase 2/3, multi-arm, multi-stage, open-label study of human leukocyte antigen (HLA)-A*02:01 negative participants with metastatic uveal melanoma (MUM) who will be randomized to receive either IDE196 + crizotinib or investigator's choice of treatment (pembrolizumab, ipilimumab + nivolumab, or dacarbazine).

DETAILED DESCRIPTION:
This study is designed as a multi-stage Phase 2 study within a Phase 3 study to evaluate the safety, tolerability, pharmacokinetics, dose-exposure relationship, and anti-tumor activity of IDE196 in combination with crizotinib compared to the comparator arm of investigator's choice of treatment (pembrolizumab, ipilimumab + nivolumab, or dacarbazine).

The Phase 2a dose optimization stage will evaluate two doses of IDE196 in combination with crizotinib compared to the comparator arm. Participants will be randomized to the three treatment arms. At the point of optimal IDE196 + crizotinib dose selection, the other dose arm will be dropped with discontinuation of enrollment to that arm. Participants receiving the IDE196 dose (in combination with crizotinib) that is not selected, will be offered the choice to remain on the same dose or change to the chosen optimal dose.

The optimal dose will be chosen to complete the Phase 2b portion. The Phase 2b part of the study will continue to enroll the chosen combination dose of IDE196 + crizotinib compared with the comparator arm. Participants will be randomized to the two treatment arms.

The Phase 3 part of the study will continue to enroll the chosen combination dose of IDE196 + crizotinib compared with the comparator arm. Participants will be randomized to the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed Metastatic Uveal Melanoma
* HLA-A*02:01 negative
* No prior systemic therapy in the metastatic or advanced setting or regional or liver-directed therapy. Ablations or surgical resection of oligometastatic disease, and neoadjuvant or adjuvant therapy is allowed
* Measurable disease per RECIST 1.1
* Able to be safely administered and absorb study therapy
* ECOG performance status 0 or 1
* Life expectancy of ≥3 months
* Adequate organ function

Exclusion Criteria:

* Previous treatment with a PKC inhibitor (including prior treatment with IDE196), an inhibitor directly targeting MET, or an inhibitor directly targeting GNAQ/11
* Concurrent malignant disease
* AEs from prior anti-cancer therapy that have not resolved to Grade ≤1
* Symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require corticosteroids
* High risk of syncope
* Known AIDS related illness or active Hep B/C
* Active adrenal insufficiency, active colitis, or active inflammatory bowel disease
* History of interstitial lung disease, active pneumonitis, or history of pneumonitis
* Active infection requiring systemic antibiotic therapy
* Use of hematopoietic colony-stimulating factors (CSF) prior to start of study drug
* Females who are pregnant or breastfeeding
* History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies
* Contraindication for treatment with investigator's choice therapies as per applicable labelling
* History of stroke within the last 6 months of the first dose of study drug
* Has any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the opinion of the investigator, would make the participant inappropriate for entry into the study, including institutionalization on the basis of an official or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by blinded independent central review (BICR) of IDE196 + Crizotinib compared to investigator's choice of treatment | Approximately 2 years
  PFS per RECIST 1.1
Overall Survival (OS) of IDE196 + Crizotinib compared to investigator's choice of treatment | Approximately 4 years
  OS from randomization to date of death due to any cause

SECONDARY OUTCOMES:
Safety of IDE196 + Crizotinib: Incidence of Adverse Events | Approximately 2 years
  Treatment emergent adverse events will be summarized by all AEs, all Grade 3-4-5 AEs, all treatment related AEs, all AEs leading to study drug modifications or discontinuations, all SAEs as measured by CTCAE V5.0
Phase 2a: Dose exposure response of IDE196 | Approximately 5 months
  Dose-exposure-response of IDE196 as measured by concentration of IDE196 in plasma
Phase 2a: Dose exposure response of Crizotinib | Approximately 5 months
  Dose-exposure-response of Crizotinib as measured by concentration of Crizotinib in plasma
Progression-Free Survival (PFS) per Investigator of IDE196 + Crizotinib compared to investigator's choice of treatment | Approximately 2 years
  PFS per RECIST 1.1
Objective Response Rate (ORR) per BICR and Investigator assessment of IDE196 + Crizotinib compared to investigator's choice of treatment | Approximately 2 years
  ORR per RECIST 1.1
Duration of Response (DOR) per BICR and Investigator assessment of IDE196 + Crizotinib compared to investigator's choice of treatment | Approximately 2 years
  DOR per RECIST 1.1
Change from baseline over time and between treatment arms in EORTC QLQ-C30 | Approximately 2 years
  Global health status and quality of life will be assessed using the EORTC QLQ-C30 questionnaire. The score range for the EORTC QLQ-C30 is from 0 to 100, with higher scores indicating better functioning and better global health status and health-related quality of life. A positive change indicates improvement.
Change from baseline over time and between treatment arms in EuroQoL (EQ)-5D-5L scores | Approximately 2 years
  General health status will be assessed using the EQ-5D,5L questionnaire, which includes five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 scoring levels, where 1 indicates a better health state (no problems) and 3 indicates a worse health state. A positive change indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Hetal Patel, MD, MSHS, CHCQM, Study Director — IDEAYA Biosciences
Locations (68):
- United States (31):
  - Honor Health, Scottsdale, Arizona
  - Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - California Pacific Medical Center (CPMC), San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - SCRI at HealthONE, Denver, Colorado
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital Atlanta, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, P.A., Burnsville, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology- DFW, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexander Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Washington
  - Queen Elizabeth Hospital, Adelaide
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Algemene Medische Oncologie UZ, Leuven
- Canada (4):
  - Cross Cancer Institute, University of Alberta, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal- CHUM, Montreal, Quebec
- France (2):
  - The Leon Berard Center, Lyon
  - Institut Curie, Paris
- Germany (5):
  - NCT Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen (AöR), Essen, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale dei Tumori Fondazione Pascale, Napoli
  - Fondazione Policlinico Gemelli IRCCS, Roma
  - AOUS Policlinico Le Scotte, Siena
- LUMC (Leids Universitair Medisch Centrum), Leiden, Netherlands
- Poland (2):
  - Ośrodek Badań Klinicznych Wczesnych Faz, Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Warsaw
- Spain (5):
  - Catalan Institute of Oncology, L'Hospitalet de Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario Valencia, Valencia
- Dermatologische Klinik, USZ Flughafen Geschoss 7 - Klinische Forschung, Zurich, Switzerland
- United Kingdom (3):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Mount Vernon Cancer Centre East & North Herts NHS Trust, Northwood